CLINICAL TRIAL: NCT02463643
Title: A Randomized, Double-Blind, Multicenter Study to Evaluate Efficacy and Safety of Z-215 Compared With Rabeprazole Sodium in the Treatment of Erosive Esophagitis
Brief Title: To Evaluate Efficacy and Safety of Z-215 in Erosive Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z215-01
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Esophagitis, Reflux
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Z-215 10 mg/day (Experimental): Drug: Z-215 10mg Drug: Z-215 Placebo Drug: Rabeprazole Sodium Placebo
  Interventions: Drug: Z-215 10mg; Drug: Z-215 Placebo; Drug: Rabeprazole Sodium Placebo
- Z-215 20 mg/day (Experimental): Drug: Z-215 20mg Drug: Z-215 Placebo Drug: Rabeprazole Sodium Placebo
  Interventions: Drug: Z-215 20mg; Drug: Z-215 Placebo; Drug: Rabeprazole Sodium Placebo
- Z-215 40 mg/day (Experimental): Drug: Z-215 20mg Drug: Z-215 20mg Drug: Rabeprazole Sodium Placebo
  Interventions: Drug: Z-215 20mg; Drug: Rabeprazole Sodium Placebo
- Rabeprazole Sodium 10 mg/day (Active Comparator): Drug: Z-215 Placebo Drug: Z-215 Placebo Drug: Rabeprazole Sodium
  Interventions: Drug: Z-215 Placebo; Drug: Rabeprazole Sodium

INTERVENTIONS:
Drug: Z-215 10mg — Z-215 10mg, capsules
  Arms: Z-215 10 mg/day
Drug: Z-215 20mg — Z-215 20mg, capsules
  Arms: Z-215 20 mg/day; Z-215 40 mg/day
Drug: Z-215 Placebo — Z-215 placebo-matching capsules
  Arms: Rabeprazole Sodium 10 mg/day; Z-215 10 mg/day; Z-215 20 mg/day
Drug: Rabeprazole Sodium — Rabeprazole Sodium 10mg tablets
  Arms: Rabeprazole Sodium 10 mg/day
Drug: Rabeprazole Sodium Placebo — Rabeprazole Sodium Placebo placebo-matching tablets
  Arms: Z-215 10 mg/day; Z-215 20 mg/day; Z-215 40 mg/day

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Z-215 (10 mg, 20 mg, 40 mg) , compared with Rabeprazole Sodium 10mg in patients with erosive esophagitis of Grade A to D as defined by the LA classification grading system.

ELIGIBILITY:
Inclusion Criteria:

* In observation period, the participant must have endoscopically confirmed erosive esophagitis of Grade A to D, as defined by the LA classification grading system, and the target number of participants who are clearly Grade C or D is 20% (96 participants) or more of the total participants.
* Outpatient (including inpatient for examination)

Exclusion Criteria:

* Participants with a previous or current history of eosinophilic esophagitis,scleroderma, esophageal stenosis, esophageal varices, Barrett's esophagus ( columnar epithelium metaplasia>=3 cm ) or high-grade dysplasia.However, participants with Schatzki's ring ( >=20mm ) are allowed to be included.
* Participants who have acute upper gastrointestinal bleeding, gastric or duodenal ulcer (mucosal defect with white coating>=3mm) within 28 days prior to observation period . Participants with above disease at endoscopy during the observation period.
* Participants with Zollinger-Ellison syndrome.Participants with suspected gastric acid hypersecretion disorders attributable to hyperparathyroidism and others.
* Participants with a previous history of surgery of esophagus,stomach or duodenum (excluding removal of benign polyp by endoscopic polypectomy) .

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Endoscopic Healing Rate Over 8 Weeks of Erosive Esophagitis | 8 weeks

SECONDARY OUTCOMES:
Endoscopic Healing Rate Over 4 Weeks of Erosive Esophagitis | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan